CLINICAL TRIAL: NCT06349811
Title: A Phase I Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetics Characteristics and Preliminary Efficacy of BL-M05D1 in Patients With Locally Advanced or Metastatic Solid Tumors
Brief Title: A Study of BL-M05D1 in Patients With Locally Advanced or Metastatic Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Sichuan Baili Pharmaceutical Co., Ltd. (Industry)
Collaborators: Baili-Bio (Chengdu) Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BL-M05D1-101
Record Dates: First submitted 2024-04-01; First posted 2024-04-05 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Locally Advanced or Metastatic Solid Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BL-M05D1 (Experimental): Participants receive BL-M05D1 as intravenous infusion for the first cycle (3 weeks). Participants with clinical benefit could receive additional treatment for more cycles. The administration will be terminated because of disease progression or intolerable toxicity occurring or other reasons.
  Interventions: Drug: BL-M05D1

INTERVENTIONS:
Drug: BL-M05D1 — Administration by intravenous infusion for a cycle of 3 weeks.

SUMMARY:
This study is an open-label, multicenter, dose-escalation, and extended-enrollment nonrandomized phase I study to evaluate the safety, tolerability, pharmacokinetic characteristics, and preliminary efficacy of BL-M05D1 in patients with locally advanced or metastatic solid tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Sign the informed consent form voluntarily and follow the protocol requirements;
2. Gender is not limited;
3. Age: ≥18 years old and ≤75 years old;
4. Expected survival time ≥3 months;
5. locally advanced or metastatic solid tumors confirmed by histopathology and/or cytology with failure or intolerance to standard treatment or no standard treatment at present;
6. Consent to provide archival tumor tissue samples or fresh tissue samples from primary or metastatic lesions within 3 years;
7. At least one measurable lesion meeting the RECIST v1.1 definition was required;
8. ECOG 0 or 1;
9. The toxicity of previous antineoplastic therapy has returned to ≤ grade 1 as defined by NCI-CTCAE v5.0;
10. No severe cardiac dysfunction, left ventricular ejection fraction ≥50%;
11. No blood transfusion, no use of cell growth factors and/or platelet-raising drugs within 14 days before screening, and the organ function level must meet the requirements;
12. Coagulation function: international normalized ratio (INR) ≤1.5, and activated partial thromboplastin time (APTT) ≤1.5ULN;
13. Urinary protein ≤2+ or ≤1000mg/24h;
14. For premenopausal women with childbearing potential, a pregnancy test must be performed within 7 days before starting treatment, serum pregnancy must be negative, and the patient must not be lactating; All enrolled patients (male or female) were advised to use adequate barrier contraception throughout the treatment cycle and for 6 months after the end of treatment.

Exclusion Criteria:

1. Chemotherapy, biological therapy, immunotherapy and other anti-tumor therapies have been used within 4 weeks or 5 half-lives before the first dose; Mitomycin and nitrosoureas were administered within 6 weeks before the first dose; Oral fluorouracil or palliative radiotherapy within 2 weeks before the first dose; Chinese patent medicine within 2 weeks before the first administration;
2. History of severe cardiovascular and cerebrovascular diseases;
3. Prolonged QT interval, complete left bundle branch block, III degree atrioventricular block, frequent and uncontrollable arrhythmia;
4. active autoimmune and inflammatory diseases;
5. other malignant tumors diagnosed within 5 years before the first dose;
6. Hypertension poorly controlled by two antihypertensive drugs;
7. had a history of ILD or a suspicion of such disease on imaging during screening; The patient was diagnosed with grade ≥1 radiation pneumonitis according to the RTOG/EORTC definition;
8. Pulmonary disease defined as grade ≥2 according to CTCAE v5.0; Pulmonary diseases lead to clinically severe respiratory function impairment;
9. patients with poor glycemic control;
10. patients with active central nervous system metastases;
11. Patients with massive or symptomatic effusions, or poorly controlled effusions;
12. Imaging examination showed that the tumor had invaded or wrapped around the chest, neck, pharynx and other large blood vessels;
13. had a history of pulmonary embolism or a thrombotic event requiring therapeutic intervention within 6 months before screening; Infusion-related thrombosis was excluded;
14. had a history of allergy to recombinant humanized antibody or human-mouse chimeric antibody or any of BL-M05D1 ingredients;
15. prior organ transplantation or allogeneic hematopoietic stem cell transplantation (Allo-HSCT);
16. The cumulative dose of anthracyclines > 360 mg/m2 in previous (new) adjuvant therapy;
17. human immunodeficiency virus antibody positive, active tuberculosis, active hepatitis B virus infection or active hepatitis C virus infection;
18. active infection requiring systemic therapy;
19. had participated in another clinical trial within 4 weeks before the first dose;
20. pregnant or lactating women;
21. The investigator did not consider it appropriate to apply other criteria for participation in the trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-04-19 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Phase Ia: Dose limiting toxicity (DLT) | Up to 21 days after the first dose
  DLTs are assessed according to NCI-CTCAE v5.0 during the first cycle and defined as occurrence of any of the toxicities in DLT definition if judged by the investigator to be possibly, probably or definitely related to study drug administration.
Phase Ia: Maximum tolerated dose (MTD) | Up to 21 days after the first dose
  MTD is defined as the highest dose level at which no more than 1 in 6 participants experienced a DLT during the first cycle .
Phase Ib: Recommended Phase II Dose (RP2D) | Up to approximately 24 months
  The RP2D is defined as the dose level chosen by the sponsor (in consultation with the investigators) for phase II study, based on safety, tolerability, efficacy, PK, and PD data collected during the dose escalation study of BL-M05D1.

SECONDARY OUTCOMES:
Treatment-Emergent Adverse Event (TEAE) | Up to approximately 24 months
  TEAE is defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally emerging, or any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a pre-existing condition during the treatment of BL-M05D1 . The type, frequency and severity of TEAE will be evaluated during the treatment of BL-M05D1.
Cmax | Up to approximately 24 months
  Maximum serum concentration (Cmax) of BL-M05D1 will be investigated.
Tmax | Up to approximately 24 months
  Time to maximum serum concentration (Tmax) of BL-M05D1 will be investigated.
T1/2 | Up to approximately 24 months
  Half-life (T1/2) of BL-M05D1 will be investigated.
AUC0-t | Up to approximately 24 months
  AUC0-t is defined as area under the serum concentration-time curve from time 0 to the time of the last measurable concentration.
CL (Clearance) | Up to approximately 24 months
  CL in the serum of BL-M05D1 per unit of time will be investigated.
Ctrough | Up to approximately 24 months
  Ctrough is defined as the lowest serum concentration of BL-M05D1 prior to the next dose will be administered.
ADA (anti-drug antibody) | Up to approximately 24 months
  Frequency of anti-BL-M05D1 antibody (ADA) will be investigated.
Phase Ib: Objective Response Rate (ORR) | Up to approximately 24 months
  ORR is defined as the percentage of participants, who has a CR (disappearance of all target lesions) or PR (at least a 30% decrease in the sum of diameters of target lesions). The percentage of participants who experiences a confirmed CR or PR is according to RECIST 1.1.
Phase Ib: Disease Control Rate (DCR) | Up to approximately 24 months
  The DCR is defined as the percentage of participants who has a CR, PR, or Stable Disease (SD: neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease [PD: at least a 20% increase in the sum of diameters of target lesions and an absolute increase of at least 5 mm. The appearance of one or more new lesions is also considered PD]).
Phase Ib: Duration of Response (DOR) | Up to approximately 24 months
  The DOR for a responder is defined as the time from the participant's initial objective response to the first date of either disease progression or death, whichever occurs first.

CONTACTS AND LOCATIONS:
Overall Officials: Lin Shen, PHD, Principal Investigator — Peking University Cancer Hospital & Institute
Locations (1):
- Beijing Cancer Hospital, Beijing, Beijing Municipality, China